CLINICAL TRIAL: NCT01417390
Title: Randomized Phase Ⅱ Trial of Induction Chemotherapy Using Gemcitabine and Cisplatin in Concurrence With Intensity-modulated Radiotherapy for Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Study of Neoadjuvant Gemcitabine and Cisplatin in Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Tao Xu, Foshan head and neck group, First People's Hospital of Foshan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FSHNG-1108
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concurrent chemoradiotherapy (Experimental): Patients receive radical radiotherapy with IMRT and cisplatin (40mg/m2) every week for six cycles during radiotherapy
  Interventions: Drug: Cisplatin
- Inductive and concurrent (Experimental): Patients receive Gemcitabine (1000mg/m2 on day 1,8) and cisplatin (20mg/m2 on day 1-4) every three weeks for two cycles before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (40mg/m2) every week for six cycles during radiotherapy.
  Interventions: Drug: Drug: Gemcitabine and cisplatin

INTERVENTIONS:
Drug: Drug: Gemcitabine and cisplatin — Patients receive Gemcitabine (1000mg/m2 on day 1,8) and cisplatin (20mg/m2 on day 1-4) every three weeks for two cycles before the radiotherapy, then receive radical radiotherapy with IMRT and cisplatin (40mg/m2) every week for six cycles during radiotherapy.
  Other Names: Gemcitabine and cisplatin
  Arms: Inductive and concurrent
Drug: Cisplatin — Patients receive radical radiotherapy and cisplatin (40mg/m2) every week for six cycles during radiotherapy
  Arms: Concurrent chemoradiotherapy

SUMMARY:
The purpose of this study is to compare induction chemotherapy (gemcitabine+cisplatin) plus concurrent chemoradiotherapy with concurrent chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma (NPC), in order to confirm the value of induction chemotherapy using gemcitabine and cisplatin in NPC patients.

DETAILED DESCRIPTION:
Patients presented with non-keratinizing NPC and stage Ⅲ-Ⅳb T3-4N1M0/TxN2-3M0 are randomly assigned to receive induction chemotherapy (gemcitabine+cisplatin) plus concurrent chemoradiotherapy (investigational arm) or concurrent chemoradiotherapy (control arm). Patients in both arms receive radical Intensity modulated radiation therapy (Trilogy, Varian), and cisplatin (40mg/m2) every weeks for six cycles during radiotherapy. Radiation is delivered to GTV at 70 Gy in 30 fractions, CTV1 at at 60 Gy in 30 fractions and CTV2 at 54 Gy in 30 fractions. Patients in the investigational arm receive gemcitabine (1000mg/m2 on day 1,8) and cisplatin (20mg/m2 on day 1-4) every three weeks for two cycles before the radiotherapy. The primary end point is response rates after radiotherapy, failure-free survival (FFS) and toxic effects and treatment compliance. Secondary end points include overall survival (OS), distant failure-free survival (D-FFS), locoregional failure-free survival (LR-FFS). All efficacy analyses are conducted in the intention-to-treat population; the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to World Health Organization (WHO 2005) histologically type).
* Karnofsky scale (KPS) > 70.
* Tumor staged is according to the 7th American Joint Commission on Cancer edition as Stage III：T1-2N2M0, T3N0-2M0 Stage IVa：T4N0-2M0 Stage IVb：Any T、N3.
* Adequate marrow: leucocyte count ≥4000/μL, hemoglobin ≥90g/L and platelet count ≥100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT)、Aspartate Aminotransferase (AST) <1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤2.5×ULN, and bilirubin ≤ULN.
* Adequate renal function: creatinine clearance ≥60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma.
* Age >60 years or <18 years.
* Treatment with palliative intent.
* Pregnancy or lactation.
* Prior radiotherapy, chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease including unstable cardiac disease, chronic hepatitis, renal disease, diabetes with poor control, and emotional disturbance.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3-year
  Failure-free survival is calculated from the date of randomization to the date of the first failure at any site.

SECONDARY OUTCOMES:
Overall survival | 3-year
  Overall survival is calculated from randomization to death from any cause.
Locoregional failure-free survival | 3-year
  the latency to the first local failure
Distant failure-free survival | 3-year
  The latency to the first remote failure
The initial response rates after treatments | 16 weeks after completion of radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Wei-wei Hong, Foshan, Guangdong, China

REFERENCES:
- [Background] He X, Ou D, Ying H, Zhu G, Hu C, Liu T. Experience with combination of cisplatin plus gemcitabine chemotherapy and intensity-modulated radiotherapy for locoregionally advanced nasopharyngeal carcinoma. Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1027-33. doi: 10.1007/s00405-011-1669-9. Epub 2011 Jun 26. Erratum In: Eur Arch Otorhinolaryngol. 2012 Mar;269(3):1035. Xiayun, He [corrected to He, Xiayun]. PMID 21706324
- [Background] Drossigk U, Hiepe T, Potzsch F, Scholz D, Tietz HJ. Stimulation of human immunodeficiency virus expression in permanent monocytic cells by Sarcocystis gigantea extract. Parasitol Res. 1998 Jun;84(6):455-8. doi: 10.1007/s004360050429. PMID 9660134
- [Background] Lowy AM, Firdaus I, Roychowdhury D, Redmond K, Howington JA, Sussman JJ, Safa M, Ahmad SA, Reed MF, Rose P, James L, Jazieh AR. A phase II study of sequential neoadjuvant gemcitabine and paclitaxel, radiation therapy with cisplatin and 5-fluorouracil and surgery in locally advanced esophageal carcinoma. Am J Clin Oncol. 2006 Dec;29(6):555-61. doi: 10.1097/01.coc.0000233997.36073.8e. PMID 17148991
- [Background] Yau TK, Lee AW, Wong DH, Yeung RM, Chan EW, Ng WT, Tong M, Soong IS. Induction chemotherapy with cisplatin and gemcitabine followed by accelerated radiotherapy and concurrent cisplatin in patients with stage IV(A-B) nasopharyngeal carcinoma. Head Neck. 2006 Oct;28(10):880-7. doi: 10.1002/hed.20421. PMID 16721741
- [Background] Chua DT, Sham JS, Au GK. Induction chemotherapy with cisplatin and gemcitabine followed by reirradiation for locally recurrent nasopharyngeal carcinoma. Am J Clin Oncol. 2005 Oct;28(5):464-71. doi: 10.1097/01.coc.0000180389.86104.68. PMID 16199985
- [Background] Benasso M, Merlano M, Sanguineti G, Corvo R, Numico G, Ricci I, Pallestrini E, Santelli A, Vitale V, Marchetti G, Rosso R. Gemcitabine, cisplatin, and radiation in advanced, unresectable squamous cell carcinoma of the head and neck: a feasibility study. Am J Clin Oncol. 2001 Dec;24(6):618-22. doi: 10.1097/00000421-200112000-00019. PMID 11801767